CLINICAL TRIAL: NCT04239261
Title: A Randomized, Placebo-Controlled, Pilot Study of Serum-Derived Bovine Immunoglobulin/Protein Isolate to Manage Mucositis in Patients Undergoing Treatment for Head, Neck, or Lung Cancer
Brief Title: Serum-derived Bovine Immunoglobulin Effect on Mucositis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment slower than anticipated
Sponsor: MercyOne Des Moines Medical Center (Other)
Responsible Party: Principal Investigator, Richard Deming, MD, Principal Investigator, MercyOne Des Moines Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HNL-MUCO
Record Dates: First submitted 2020-01-14; First posted 2020-01-27 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Mucositis
MeSH Terms: conditions — Mucositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nutritional therapy (Active Comparator): Serum-derived bovine immunoglobulin/protein isolate (SBI) 10.0 grams once daily
  Interventions: Dietary Supplement: SBI
- Placebo (Placebo Comparator): Hydrolyzed gelatin 10.0 grams once daily
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: SBI — Serum-derived Bovine immunoglobulin/protein isolate 10.0 g once daily
  Arms: Nutritional therapy
Dietary Supplement: Placebo — Hydrolyzed gelatin 10.0 g once daily
  Arms: Placebo

SUMMARY:
The purpose of this cancer control clinical research study is to evaluate whether nutritional therapy with Serum-derived bovine immunoglobulin/protein isolate (SBI) might reduce mucositis (a condition caused by cancer treatment involving mouth sores, pain and/or bleeding that may cause difficulty eating), improve nutritional status and lessen the symptoms associated with chemo-radiation therapy which may result in quality of life (QOL) improvements during the prescribed treatment for cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained and signed
2. Male or female at least 18 years of age
3. Diagnosed with head, neck, or lung cancer and scheduled to undergo combined chemo-radiation therapy
4. Diagnosed with head, neck, or lung cancer with disease stage within the criteria described in 4.0 Staging Criteria
5. Not experiencing diarrhea during the 5 days preceding enrollment, as defined by having less than two unformed bowel movements per day or loose (mushy) or watery stools in the 5 days preceding enrollment.
6. Not currently taking anti-diarrheal medications (prescription or over the counter).
7. Agrees and is able to take the investigational products or placebo starting from the day of enrollment (approximately 7-14 days prior to beginning chemo-radiation therapy) through 6-7 weeks of chemo-radiation therapy (for a total of 8-9 weeks).

Exclusion Criteria:

1. History of uncontrolled diarrhea during screening.
2. History of Irritable Bowel Syndrome with Diarrhea with a normal pattern of more than three bowel movements in a 24 hour period.
3. History of inflammatory bowel disease: ulcerative colitis, Crohn's disease, or microscopic colitis.
4. History of active infectious diarrhea and receiving therapy within 10 days of the first dose of study drug or placebo.
5. Known allergy or intolerance to beef or soy or any ingredient used in the product
6. History of concurrent intensive chemotherapy within 10 days of the first scheduled dose of study drug or placebo.
7. Gastrointestinal surgery or bowel resection that could affect study product absorption (this does not include cholecystectomy or appendectomy).
8. Unable to comply with the protocol requirements.
9. Any condition that in the opinion of the Investigator might interfere with the study objective.
10. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Development of Oral Mucositis during ChemoRadiation Treatment | Baseline and Up to approximately 90 days after randomization
  CTCAE version 5 will be used to determine adverse event grade of mucositis, if applicable

SECONDARY OUTCOMES:
Development of Dysphagia during ChemoRadiation Treatment | Baseline and Up to approximately 90 days after randomization
  CTCAE version 5 will be used to determine advent grade of dysphagia, if applicable
Change in Bowel Movements | Baseline and Up to approximately 90 days after randomization
  Stool Diary Card will be completed by patient to document consistency, ease and completeness

CONTACTS AND LOCATIONS:
Overall Officials: Richard Deming, MD, Principal Investigator — MercyOne Des Moines Medical Center
Locations (1):
- MercyOne Des Moines Medical Center, Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: No